CLINICAL TRIAL: NCT05132647
Title: Circular Timed Up and Go (cTUG) Test for Assessing Balance and Falls Risk Among Individuals With Cerebellar Ataxia: Development and Validation
Brief Title: Circular Timed Up and Go (cTUG) for Ataxia: Development and Validation
Acronym: cTUG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: P0030822
Record Dates: First submitted 2021-10-17; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Cerebellar Ataxia; Healthy Adults
Keywords: cerebellar ataxia,; falls risk,; outcome measures; falls prevention
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebellar ataxia and Healthy adults: We will not administer any intervention to the patients in this study

SUMMARY:
Cerebellar ataxia (CA) is a collection of signs and symptoms caused by cerebellar dysfunction, which can be the result of different disease processes including hereditary and acquired conditions. High incidence of falls is reported in people with CA due to poor balance while walking. Therefore, it is crucial to assess the balance of people with CA to identify potential fallers. There are some clinical tests commonly used for assessing the balance of people with CA, including both generic measures of balance and ataxia-specific rating scales. The current best balance outcome measures for CA includes Berg Balance Scale (BBS), Timed Up and Go test (TUG), and the balance related items in Scale for the assessment and rating of ataxia (SARA). TUG is commonly used in clinical settings for the assessment of mobility and fall risk of individuals. However, a study done by Winser et. al (2017) found that the correlation between TUG and ataxia rating scales (SARA and ICARS) is only moderate. This indicates that the gait speed and functional mobility findings of TUG might not truly reflect the balance deficits of CA. Therefore, our study will develop a modified TUG for the assessment of balance in people with CA. Circular TUG (cTUG) is a modified version of the standard TUG. cTUG is an equilibrium test that challenges subjects' ability to maintain balance in response to the constant change in direction of walking. In cTUG, the subject walks a semi-circular pathway instead of a straight line. Walking in a circular pathway targets at challenging the coordination of people with CA as walking in a circle requires constant change in directions and correction after feedback. It is speculated that the cTUG will have better accuracy in predicting the balance and falls risk among people with CA. We will target at recruiting 30 healthy volunteers and 30 individuals with cerebellar ataxia. Besides the cTUG we will also assess disease severity of ataxia using the Scale for the Assessment and Rating of Ataxia (SARA), balance using the Berg Balance Scale, Timed Up and Go test, Sensory Organization test, Limits of Stability test and functional independence using the Barthel Index. For validation of the cTUG, two types of reliability will be examined, including intra-rater reliability and interrater reliability and four types of validity will be assessed, including concurrent validity, convergent validity, discriminant validity, and external validity.

DETAILED DESCRIPTION:
Background What is Cerebella ataxia (CA)? Cerebellar ataxia (CA) is a collection of signs and symptoms caused by cerebellar dysfunction, which can be the result of different disease processes including hereditary and acquired conditions (Hadjivassiliou et al., 2017).

Common clinical presentation of CA patients includes balance and gait dysfunction, dysmetria, dyssynergia, dysarthria and dysdiadochokinesia (Diener & Dichgans, 1992). People with CA usually walks with increased step width, increased foot rotation angles and reduced cadence, which is related to impaired balance (Stolze et al., 2002). Marsden & Harris (2011) suggested that the high incidence of falls in people with CA may be related to their poor balance in walking. Therefore, it is crucial to assess the balance of people with CA to identify potential fallers.

Current balance assessments and drawbacks of TUG There are some clinical tests commonly used for assessing the balance of people with CA, including both generic measures of balance and ataxia-specific rating scales. The current best balance outcome measures for CA includes Berge Balance Scale (BBS), Timed Up and Go test (TUG), and the balance related items in Scale for the assessment and rating of ataxia (SARA) (Winser et al., 2015). TUG is commonly used in clinical settings for the assessment of mobility and fall risk of individuals (Dawson et al., 2018). However, a study done by Winser et. al (2017) found that the correlation between TUG and ataxia rating scales (SARA and ICARS) is only moderate. This indicates that the gait speed and functional mobility findings of TUG might not truly reflect the balance deficits of CA. Therefore, in order to bridge this gap, our study will develop a modified TUG for the assessment of balance in people with CA. The specific objectives of this study will be to examine the reliability, validity of the modified TUG for identifying the balance and fall risk of cerebellar ataxia patients.

Circular TUG: A modification that might suit CA Circular TUG (cTUG) is a modified version of the standard TUG. cTUG is an equilibrium test that challenges subjects' ability to maintain balance in response to constant change in direction of walking. In standard TUG, the person gets up from an armchair, walks three meters in a straight pathway, then turn 180 degrees and walks back to the chair to sit down (Podsiadlo & Richardson, 1991b). However, in cTUG, the subject walks a semi-circular pathway instead of a straight line. Walking in a circular pathway targets at challenging the coordination of people with CA as walking in a circle requires constant change in directions and correction after feedback (Goodworth et al., 2012). Moreover, walking in a circle is more difficult for patients with CA as it increases the role of the cerebellum for trunk and foot control during curvilinear locomotion (Goodworth et al., 2012). Therefore, it is speculated that the cTUG will have better accuracy in predicting the balance and falls risk among people with CA.

Objectives and hypothesis The overall aim of this study is to develop and test the psychometric properties of the cTUG in assessing balance and falls risk prediction among individuals with cerebellar ataxia and age-matched healthy volunteers. To address this objective, we have the following specific objectives.

1. Develop the cTUG and record the normative scores of the newly developed scale among healthy volunteers and mean scores among individuals with cerebellar ataxia.
2. Examine the test-retest, inter-rater and intra-rater reliability of the cTUG among healthy volunteers and individuals with cerebellar ataxia.
3. Examine the concurrent validity, convergent validity, discriminant validity, and external validity of the cTUG among individuals with cerebellar ataxia.

For validity, concurrent validity, convergent validity, discriminant validity, and external validity will be assessed. Based on the findings of a previous study that reported a moderate negative correlation (-0.62) between standard TUG and Berg Balance scale (BBS) (Cattaneo et al., 2006), we hypothesize a moderate to strong negative correlation between cTUG and BBS.

Moreover, based on the findings of a previous study that reported a moderate positive correlation (0.584) between standard TUG and Scale for the Assessment and Rating of Ataxia (SARA) (Choi et al., 2018), we hypothesize a moderate to strong positive correlation between cTUG and the balance component SARA.

In addition, based on the findings of a previous study that reported a positive correlation between TUG and Modified Clinical Test of Sensory Organization and Balance (m-CTSIB) and a negative correlation between TUG and Limit of Stability (LOS) (Dawson et al., 2018), we hypothesize a positive correlation between cTUG and Sensory Organization Test (SOT), and a negative correlation between cTUG and LOS.

Besides, based on the findings of a previous study that reported a moderate negative correlation (-0.78) between standard TUG and Barthel Index (BI) (Podsiadlo & Richardson, 1991b), we hypothesize a moderate negative correlation between cTUG and BI.

For reliability, intra-rater reliability and inter-rater reliability will be assessed. Repeat assessment by the same investigator will be used to estimate intra-rater reliability and repeat assessments by 2 different investigators will be used to estimate inter-rater reliability. All the assessments will be completed on the same day with each assessment conducted with 1 hour rest period.

Ethics will be obtained through the Human Subjects Ethics Sub-committee of the Hong Kong Polytechnic University and trial registration will be done through the Clinical Trials Registry. Participants with a confirmed diagnosis of CA of any or unknown cause will be recruited through the Hong Kong Spinocerebellar Ataxia Association (HKSCAA) and one group of age-matched healthy volunteers will be recruited from the Hong Kong PolyU campus. We will post advertisement flyers at the HK PolyU campus and at the HKSCAA for recruiting potential participants. In addition, for recruiting participants with cerebellar ataxia, an advertisement flyer will be posted on the monthly newsletter of the HKSCAA. The specific criteria for recruitment are reported elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* CA patients (hereditary, degenerative or acquired underlying cause)
* ambulatory
* age 18-65
* able to walk independently with or without assistive walking device for at least 10m

Exclusion Criteria:

* CA patients who require hand held support during walking
* CA patients with severe visual impairment
* Expanded Disability Status Scale (EDSS) score >6.5
* Refuse to reveal personal information
* CA patients with other associated neurological conditions that does not result in ataxia features
* Poor cognition or unable to follow the instructions

Healthy adults: Both genders aged 18 to 65 who are ambulant with or without assistive device for walking.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants with a confirmed diagnosis of cerebellar ataxia secondary to sporadic, degenerative or acquired cause will be considered.
  Healthy adults are those who are ambulant with or without the use of a walking assistive device.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Circular TUG (cTUG) | Baseline (T1), Day 1 (T2) and Day 1 (T3)
  Circular TUG (cTUG) is a modified version of the standard TUG. cTUG is an equilibrium test that challenges subjects' ability to maintain balance in response to constant change in direction of walking. In standard TUG, the person gets up from an armchair, walks three meters in a straight pathway, then turn 180 degrees and walks back to the chair to sit down (Podsiadlo & Richardson, 1991b). However, in cTUG, the subject walks a semi-circular pathway instead of a straight line.

SECONDARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | Assessment 1 day 1
  The Scale for the Assessment and Rating of Ataxia (SARA) is a measure to assess the severity of cerebellar ataxia. There are total of 8 items: gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movement and heel-shin slide. The total score ranges from 0 to 40, which indicates no ataxia to severe ataxia. SARA has high inter-rater reliability (ICC = 0.98) and high test-retest reliability (ICC = 0.90) in assessing cerebellar ataxia patients. Internal consistency is high as indicated by Cronbach's α of 0.94 (Schmitz-Hubsch et al., 2006).
Berg Balance Scale (BBS) | Assessment 1 day 1
  Berg Balance Scale (BBS) measures the ability in maintaining balance during tasks. The scale consists of 14 items, requiring patients to maintain different positions for specific durations. Each item is rated from 0 to 4, from lowest ability to highest ability. The time and quality in maintaining positions are assessed. The maximum score is 56. Score of less than 45 indicates higher fall risk (Katherine et al., 1992). The test has good inter-rater reliability (ICC = 0.96) and high test-retest reliability (ICC = 0.94) (Cattaneo et al., 2007).
The timed up and go test | Assessment 1 on Day 1, Assessment 2 on day 1 and Assessment 3 on day 2
  The timed up and go test is a test to quantify the functional mobility by balance, gait speed and functional capacity. The subject is timed while asked to stand up from a chair, walks 3 meters, turns and walks back and sits down again. Those who takes more than 30 seconds to complete the test are considered having poor balance and require assistance for many mobility tasks. Those completed the test in less than 10 seconds are considered very independent in mobility tasks (Podsiadlo & Richardson, 1991a).
Sensory organization test (SOT) | Assessment 1 day 1
  Sensory organization test (SOT) is an objective evaluation on postural stability under different sensory conditions. The test is performed with the Bertec System. Subjects are challenged to stand unsupported under six sensory scenarios, with different visual, somatosensory and vestibular inputs. There are three trials lasting for 20 seconds in each scenario. Equilibrium score in each scenario and the composite equilibrium score are assessed. The equilibrium score provides quantitative evaluation on subjects' postural sway under different sensory conditions. Composite equilibrium score shows subjects' average performance over the trials. The score of subjects is compared to the normative data in the software database. Results falling outside normal value indicates abnormal sway and shows difficulty in incorporating sensory information for balance control. (Bertec corporation, 2014).
Limit of Stability (LOS) | Assessment 1 day 1
  Limit of Stability (LOS) is an objective balance assessment by assessing the ability to displace centre of gravity in different directions without losing balance. The test is performed with the Bertec System. Subjects are assessed in eight directions and their centre of gravity is traced during movement. The directional control (DCL), reaction time (RT) and maximum excursion (MXE) are assessed. Directional control is the measurement of how much subjects move towards the target direction. Reaction time is the time taken for subjects to respond to the command of moving towards the target. Maximum excursion is measurement of the extent that subjects lean during trials. The score of subjects is compared to the normative data in the software database. Result falling outside the normal value indicates restricted stability limit and an increased risk of falling. (Bertec corporation, 2014).
Barthel Index | Assessment 1 day 1
  The Barthel index (BI) is an ordinal scale for measuring performance in activities of daily living (ADL). There are a total of 10 variables under ADL and mobility, each values a given number of points. Higher points indicate a greater degree of independence (O'Sullivan et al., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Winser, PhD, Principal Investigator — The Hong Kong Polytechnic Universit
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The patients' personnel identification will be masked. the scores will be made available for the publisher using an anonymous ID for each participant. Personnel identifiers such as photos or names will be identified in public forums including conference presentations.